CLINICAL TRIAL: NCT03313375
Title: Postexercise Hemodynamics Compared in Obese and Non-Obese Subjects After Aerobic Interval Training
Brief Title: Continuous vs Aerobic Postexercise Hypotension
Acronym: CAPER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding and personnel
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Siddhartha Angadi, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ASU-STUDY00006782
Record Dates: First submitted 2017-10-05; First posted 2017-10-18 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Postexercise Hypotension
Keywords: hemodynamics; exercise
MeSH Terms: conditions — Post-Exercise Hypotension; Motor Activity

STUDY DESIGN:
Intervention Model Description: Subjects will have a randomized order of treatment (exercise bouts). Each subject will complete all three (control, cont. exercise, aerobic interval), but in a randomized order.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Subjects will have no intervention. They will be resting in a chair for the entire length of the visit (4-5 hours) where blood pressure will be taken every 10 min, while other non-invasive cardiac measures are taken (I.E. Cardiac output, systemic vascular resistance, heart rate variability).
- Continuous exercise (Active Comparator): Subjects will be asked to perform a 45 min exercise bout. After a warmup, the exercise will be 30 minutes at a continuous level. After the exercise period subject will remain in the lab and blood pressure will be measured every 10 minutes for the remainder of the visit (4 hours) while other non-invasive cardiac measures are taken continuously as discussed above.
  Interventions: Other: Continuous Exercise
- Aerobic Interval Exercise (Experimental): Subjects will be asked to complete a 43 minute exercise session. After a warmup period, the subjects will complete a 4x4 protocol in that they will alternate 4, 4 minute higher intensity exercise bouts with 3, 3 minute lower intensity bouts. After the exercise, subjects will remain in the lab and blood pressure will be measured every 10 minutes for 4 hours, while other non-invasive cardiac measures are taken continuously as discussed above.
  Interventions: Other: Aerobic Interval Exercise

INTERVENTIONS:
Other: Continuous Exercise — Subjects will be asked to perform a 45 min exercise bout. 10 minutes will be a warmup (at a work rate associated with 50% heart rate max), 30 minutes at a wattage that elicits 75-80% heart rate max, and a 5 minute cool down period, returning them to approximately 50% heart rate max.
  Other Names: CE
  Arms: Continuous exercise
Other: Aerobic Interval Exercise — Subjects will be asked to complete a 43 minute exercise session. To warm up, subjects will cycle at a work rate associated with 50% HRmax for 10 minutes. Wattage will then increase and subjects will do four 4-minute intervals at a work rate associated with 90%-95% HRmax, separated by 3 minutes of active recovery at a work rate associated with 50% HRmax. Subjects will be given a 5-minute cool-down period at a work rate associated with 50% HRmax.
  Other Names: AIE
  Arms: Aerobic Interval Exercise

SUMMARY:
This study examines the effect of obesity and gender on postexercise hypotension with three different randomized exercise protocols or varying intensity. Subjects will be separated into obese and non-obese groups and then further by gender. From there, they will be put through a control, continuous exercise bout, and aerobic interval bout of exercise in a randomized order over three visits. Post exercise blood pressure, as well as other non-invasive cardiac measures will be taken over a 4 hour period.

DETAILED DESCRIPTION:
Suboptimal blood pressure, defined as >115/75 mmHg by meta-analysis, exhibits a positive relationship with cardiovascular disease, and is the leading attributable risk factor for death. Research has illustrated that even blood pressure (BP) below the hypertensive levels can contribute to increased vascular mortality. It has been demonstrated that for incremental increases in blood pressure (every 20 mmHg systolic or 10 mmHg diastolic) there is a twofold increase in cardiovascular disease risk. However, mounting evidence suggests that increased fitness and physical activity4 may attenuate the typical age related increase in BP to hypertensive levels. Exercise has been recommended as the first line of treatment in prehypertension and suboptimal BP, and a single bout of exercise (as short at 10 min) has been shown to lower BP for up to 12 hours post. It is this extended bout of postexercise hypotension (PEH) that is thought to contribute to the anti-hypertensive effects of exercise.

PEH is well documented in lean and overweight individuals, but there is limited data on PEH in obese populations of both genders. Well characterized for lean and overweight individuals matched for BP, how obese men and women react postexercise is largely unknown and undefined. Only a few published studies exist. A recent meta-analysis examined PEH, but only included subjects with a body mass index of < 31 kg/m2. Only one study to date included exclusively obese subjects (all women), but the authors only demonstrated a PEH 10 min postexercise. To date, we are aware of no published data examining BP matched PEH in centrally obese men and women to that of non-obese men and women.

Exercise intensity has been shown to play a role in PEH as well. Data from this lab has demonstrated that short duration, high intensity exercise (aerobic interval exercise -AIE) was able to stimulate a greater duration of PEH when compared to that of a longer duration, moderate intensity exercise (continuous exercise- CE) or even sprint like training. One recently published study examines the effects on AIE training of young, obese women. No significant PEH was found after one hour, however, this time period may not have been long enough to see a significant change in PEH, hence why we are proposing a longer postexercise measurement period.

The mechanism for which PEH occurs is unclear. It is thought to be from structural, neurohormonal, and vascular effects of exercise, however, how these variables effect PEH in obese vs non-obese populations has not been studied directly. Using non-invasive methods such as heart rate variability (HRV), cardiac output (CO), and systemic vascular resistance (SRV) will assist us in creating a better idea of the mechanism that which PEH occurs, and any clinical difference central obesity has on these factors. A prior study from this lab found that obese subjects had a heterogeneous response in CO and SVR (increased cardiac output and augmented SVR) when compared to that of non-obese matched subjects, but once more these subjects were only evaluated for 1 hour postexercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, inactive (defined as less than 60 min of moderate to vigorous physical activity per week)
* Men (age 18-45) and non-pregnant women (age 18-55)
* Normal BMI and waist circumference (18.5- 24.5 kg/m2 and waist <94 cm ) OR obese (BMI > 30kg/m2 and waist >94 cm).
* normotensive or prehypertensive blood pressure (SBP <140 and DBP <90) according to JNC guidelines.

Exclusion Criteria:

* Subjects over age (men >45, women > 55)
* Subjects who register more than 60 minutes/week of moderate-to-vigorous physical activity via accelerometer
* Subjects who classify as hypertensive (SBP >140 or DBP >90)
* Subjects who answer positively (i.e. yes) on The Physical Activity Readiness Questionnaire (PAR-Q).
* Subjects with known cardiovascular, pulmonary, renal, or metabolic disease, or are having symptoms of these disease will be excluded, following current American College of Sports Medicine guidelines (ACSM).
* Current smokers
* Pregnant women
* Anyone with contraindications to vigorous exercise will be excluded from the study. -Subjects on medications used for the treatment of symptomatic cardiovascular disease will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Postexercise Blood pressure | Postexercise- every ten minutes for four hours post exercise session
  Central and peripheral blood pressure (systolic and diastolic) taken via Oscar 2 device.

SECONDARY OUTCOMES:
Heart Rate Variability | until study completion- up to 2 years
  Heart rate variability (taken via polar monitor)
Cardiac Output- non-invasive | until study completion- up to 2 years
  Non-invasive: taken via physioflow device
Systemic Vascular Resistance | until study completion- up to 2 years
  Non-Invasive: Taken via physioflow device

CONTACTS AND LOCATIONS:
Overall Officials: Siddhartha Angadi, PhD, Principal Investigator — Professor
Locations (2):
- United States (2):
  - Arizona Biocollaborative Building- Healthy Lifestyle research labratory, Phoenix, Arizona
  - Arizona Biomedical Collaborative 1, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prospective Studies Collaboration; Lewington S, Whitlock G, Clarke R, Sherliker P, Emberson J, Halsey J, Qizilbash N, Peto R, Collins R. Blood cholesterol and vascular mortality by age, sex, and blood pressure: a meta-analysis of individual data from 61 prospective studies with 55,000 vascular deaths. Lancet. 2007 Dec 1;370(9602):1829-39. doi: 10.1016/S0140-6736(07)61778-4. PMID 18061058
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Background] Faselis C, Doumas M, Kokkinos JP, Panagiotakos D, Kheirbek R, Sheriff HM, Hare K, Papademetriou V, Fletcher R, Kokkinos P. Exercise capacity and progression from prehypertension to hypertension. Hypertension. 2012 Aug;60(2):333-8. doi: 10.1161/HYPERTENSIONAHA.112.196493. Epub 2012 Jul 2. PMID 22753224
- [Background] Pescatello LS, Franklin BA, Fagard R, Farquhar WB, Kelley GA, Ray CA; American College of Sports Medicine. American College of Sports Medicine position stand. Exercise and hypertension. Med Sci Sports Exerc. 2004 Mar;36(3):533-53. doi: 10.1249/01.mss.0000115224.88514.3a. PMID 15076798
- [Background] Angadi SS, Weltman A, Watson-Winfield D, Weltman J, Frick K, Patrie J, Gaesser GA. Effect of fractionized vs continuous, single-session exercise on blood pressure in adults. J Hum Hypertens. 2010 Apr;24(4):300-2. doi: 10.1038/jhh.2009.110. Epub 2010 Jan 14. No abstract available. PMID 20072145
- [Background] Pescatello LS, Kulikowich JM. The aftereffects of dynamic exercise on ambulatory blood pressure. Med Sci Sports Exerc. 2001 Nov;33(11):1855-61. doi: 10.1097/00005768-200111000-00009. PMID 11689735
- [Background] Hamer M, Boutcher SH. Impact of moderate overweight and body composition on postexercise hemodynamic responses in healthy men. J Hum Hypertens. 2006 Aug;20(8):612-7. doi: 10.1038/sj.jhh.1002035. Epub 2006 Apr 20. PMID 16625235
- [Background] Angadi SS, Bhammar DM, Gaesser GA. Postexercise Hypotension After Continuous, Aerobic Interval, and Sprint Interval Exercise. J Strength Cond Res. 2015 Oct;29(10):2888-93. doi: 10.1519/JSC.0000000000000939. PMID 25785706
- [Background] Figueroa A, Baynard T, Fernhall B, Carhart R, Kanaley JA. Endurance training improves post-exercise cardiac autonomic modulation in obese women with and without type 2 diabetes. Eur J Appl Physiol. 2007 Jul;100(4):437-44. doi: 10.1007/s00421-007-0446-3. Epub 2007 Apr 4. PMID 17406886
- [Background] Liu S, Goodman J, Nolan R, Lacombe S, Thomas SG. Blood pressure responses to acute and chronic exercise are related in prehypertension. Med Sci Sports Exerc. 2012 Sep;44(9):1644-52. doi: 10.1249/MSS.0b013e31825408fb. PMID 22899388
- [Background] Carpio-Rivera E, Moncada-Jimenez J, Salazar-Rojas W, Solera-Herrera A. Acute Effects of Exercise on Blood Pressure: A Meta-Analytic Investigation. Arq Bras Cardiol. 2016 May;106(5):422-33. doi: 10.5935/abc.20160064. Epub 2016 May 6. PMID 27168471
- [Background] Bonsu B, Terblanche E. The training and detraining effect of high-intensity interval training on post-exercise hypotension in young overweight/obese women. Eur J Appl Physiol. 2016 Jan;116(1):77-84. doi: 10.1007/s00421-015-3224-7. Epub 2015 Aug 21. PMID 26293124